CLINICAL TRIAL: NCT06519747
Title: Enhanced DETECTion of PeriOperative Atrial Fibrillation After Noncardiac Surgery with Continuous Electrocardiographic Monitoring
Brief Title: DETECTion of PeriOperative Atrial Fibrillation After Noncardiac Surgery
Acronym: DETECT-POAF
Status: Recruiting | Type: Observational
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-DETECTPOAF
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Cardiac monitoring
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: Participants will receive up to 14 days of continuous cardiac monitoring
  Interventions: Device: Cardiac monitoring device

INTERVENTIONS:
Device: Cardiac monitoring device — Portable, up to 14 days of monitoring

SUMMARY:
This is a multicentre prospective cohort study where patients will receive up to 14 days of continuous ECG monitoring by wearing a portable monitoring device, starting within 72 hours after noncardiac surgery.

DETAILED DESCRIPTION:
POAF commonly occurs after noncardiac surgery and is associated with adverse long-term outcomes. Despite this, patients with POAF are routinely being missed during clinical practice. Continuous ECG monitoring has the potential to enhance POAF detection and improve clinical care in affected patients. Based on this background, the DETECT-POAF study will determine the incidence of clinically important POAF in those receiving up to 14 days of continuous ECG monitoring within 35 days after noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Had undergone noncardiac surgery within the past 72 hours and requiring, or expected to require, at least one of the following:

   * an overnight hospital admission after surgery
   * day surgery that would result in a large enough physiological insult to be able to cause POAF. Procedures excluded include those that are conducted using local anesthesia alone, are less than 30 minutes in duration, and/or are judged to be of low physiologic insult by the local investigator.
2. Have one of the following high-risk criteria;

   * age 55-64 years, and having either established cardiovascular disease, recent major vascular surgery, a CHA2DS2-VASc score ≥3, or an elevated postoperative troponin level;
   * age 65-74 years, and having either established cardiovascular disease, recent major vascular surgery, a CHA2DS2-VASc score ≥2, or an elevated postoperative troponin level; or
   * age ≥75 years;
3. Provide written informed consent to participate.

Exclusion Criteria:

1. History of documented chronic (i.e., non-transient) AF before noncardiac surgery;
2. Need for long-term systemic anticoagulation;
3. Ongoing need for long-term dual antiplatelet treatment;
4. Contraindication to oral anticoagulation;
5. Severe renal insufficiency;
6. Severe liver cirrhosis;
7. Acute stroke in the past 14 days;
8. Underwent cardiac surgery in the past 35 days;
9. History of nontraumatic intracranial, intraocular, or spinal bleeding;
10. Hemorrhagic disorder or bleeding diathesis;
11. Known life expectancy <1 year due to concomitant disease;
12. Women who are pregnant, breastfeeding, or of childbearing potential not taking effective contraception;
13. Expected to be non-compliant with follow-up and/or device use;
14. Known contact allergy to monitoring device and/or its peripheral components;
15. Previously enrolled in DETECT-POAF.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have undergone noncardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically important post-operative atrial fibrillation/atrial flutter | Within 35 days of non-cardiac surgery
  The primary outcome is clinically important POAF, defined as:
  1. Atrial fibrillation (AF) documented by a 12-lead ECG;
  2. Confirmed AF (e.g., rhythm strip) that results in symptoms of angina, heart failure, or symptomatic hypotension;
  3. Confirmed AF that requires treatment with a rate controlling drug, antiarrhythmic drug, or electrical cardioversion; or,
  4. Confirmed continuous AF episode with a minimum duration of 1 hour.

SECONDARY OUTCOMES:
Incidence of sustained ventricular arrhythmia | Within 35 days of non-cardiac surgery
Incidence of sinus node dysfunction | Within 35 days of non-cardiac surgery
Incidence of high-grade atrioventricular block | Within 35 days of non-cardiac surgery
Incidence of death | Within 35 days of non-cardiac surgery
Incidence of clinically important post-operative atrial fibrillation/atrial flutter | Within 14 days of continuous cardiac monitoring
Incidence of clinically important post-operative atrial fibrillation/atrial flutter detected by clinical monitoring only | Within 35 days of non-cardiac surgery
Incidence of clinically important post-operative atrial fibrillation/atrial flutter define with minimum duration of 6 minutes | Within 35 days of non-cardiac surgery
Incidence of clinically important post-operative atrial fibrillation/atrial flutter detected by study device monitoring only | Within 35 days of non-cardiac surgery
Proportion of participants meeting eligibility criteria for ASPIRE-AF study | Within 35 days of non-cardiac surgery
Multivariate odds ratio of risk factors associated with the occurrence of clinically important POAF | Within 35 days of non-cardiac surgery
  A multivariate logistic regression analysis of age, sex, surgical urgency, type of surgery, vascular disease, chronic kidney disease, and heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: David Conen, MD, MPH, Principal Investigator — Population Health Research Institute; Michael K Wang, MD, Principal Investigator — Population Health Research Institute
Locations (6):
- Canada (6):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Niagara Health System - St. Catharine's Site, St. Catharines, Ontario
  - Hôpital Fleurimont du Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No